CLINICAL TRIAL: NCT02644213
Title: Evaluation of Physical and Cognitive Performance After Simulated Road March Combines Physical and Cognitive Load Using a Virtual Reality Environment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: SHEBA-15-2664-OF-CTIL
Record Dates: First submitted 2015-12-23; First posted 2015-12-31 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: Physical Examination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- research arm (Experimental): 12 young, healthy civilian volunteers will participate in this study. The experiment will take place in a dome room.
  The experiment will be performed according to the protocol of using CAREN and MOTEK systems:
  1. CAREN high (Computer Assisted Rehabilitation Environment) which screens virtual scene in the dome.
  2. MOTEK (Motek Medical©, the Netherlands) which is a two track treadmill (for each leg) placed on a rotatable platform.
  each subject will undergo the same experiment protocol.
  Interventions: Other: protocol of using CAREN and MOTEK systems

INTERVENTIONS:
Other: protocol of using CAREN and MOTEK systems — The subjects will perform randomly 3 experimental days (at least weak between one to another):
  * simulated road march using a virtual reality environment without additional load
  * simulated road march using a virtual reality environment which combines cognitive load during the road march. Cognitive tasks for example: navigation, identification and remembering cars/aircraft.
  * without physical or cognitive load (without march, waiting between performance evaluations) as control.

SUMMARY:
The aim of the research is to evaluate the influence of physical and cognitive load as pre-mission activity on the soldier's physical and cognitive performance, in compare to physical load alone.

In order to do so, 12 healthy subjects will perform stimulated road march using a virtual reality environment combined with cognitive load and without, and their physical and cognitive performance will be evaluated by tests before and after.

DETAILED DESCRIPTION:
12 young, healthy civilian volunteers will participate in this study. After reading and signing an informed consent form, all subjects will undergo medical examination which includes ECG, anthropometric measurements and Vo2max test.

Afterwards, the subjects will perform randomly 3 experimental days, each consist of physical and cognitive performance evaluation before and after simulated road march using a virtual reality environment; once without additional load, once combining cognitive load during the road march, and once without physical load (without march, waiting between evaluations) as control.

The experiment will take place in a dome room, and the systems being used are:

1. CAREN high (Computer Assisted Rehabilitation Environment) which screens virtual scene in the dome.
2. MOTEK (Motek Medical©, the Netherlands) which is a two track treadmill (for each leg) placed on a rotatable platform.

cognitive tasks for example: navigation, identification and remembering cars/aircraft.

Physical and cognitive performance will be evaluated at each experimental day, before and after performing the protocol. at the end of the march, cognitive performance will be evaluated by validated tests on laptop (SYNWIN activity research services) and executive function evaluation based on Trail Making Test (TMT), afterwards, Physical performance will be evaluated by HRV and time to exhaustion test (30 min after the end of cognitive tests).

ELIGIBILITY:
Inclusion Criteria:

* aged 18-30
* healthy civilians volunteers
* with no background illnesses
* with history of combat unit service in the IDF.
* fit to perform 10 Km moderate march while carrying load.

Exclusion Criteria:

* The existence or suspicion of existing cardiac or respiratory disease.
* Hypertension.
* Diabetes.
* Any muscles or skeleton condition.
* Any hormonal disease or any other chronic illness that may inhibit participation in the experiment.
* Infectious disease 3 days prior to the experiment.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
cognitive performance (composite) | 3 experimental days
  grade will be calculated according to the subject's performance in the computerized tests (SYNWIN activity research services) at the virtual reality environment . performance evaluation is based on the parameters: concentration, memory, visual perception, data processing capability, response time and multitasking.
executive function | 3 experimental days
  executive function will be evaluated based on the validated Trail Making Test (TMT).

SECONDARY OUTCOMES:
lactic acid | 3 experimental days
  lactic acid is a marker for anaerobic effort evaluating, lactic acid level is assessed from blood drop (finger sting) using lactate scout analyzer. lactic acid will be measured before and after time to exhaustion test.
heart rate variability | 3 experimental days
  HRV will be measured during rest and effort using a wearable heart rate monitor (Polar® sensor and heart rate monitor watch).

CONTACTS AND LOCATIONS:
Overall Officials: Ofir Frenkel, M.D, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba medical center, Tel Litwinsky, Ramat- Gan, Israel